CLINICAL TRIAL: NCT02944513
Title: Efficacy of the Quell Wearable Device for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Robert N. Jamison, PhD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002172
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Subjects will receive the Quell device
  Interventions: Device: Quell
- Control (No Intervention): Subjects will not receive the Quell device

INTERVENTIONS:
Device: Quell
  Arms: Experimental

SUMMARY:
This is a 1-year trial designed to gather information about the use of the Quell for persons with chronic musculoskeletal low back pain.

DETAILED DESCRIPTION:
Research Objectives: This is a 1-year trial designed to gather information about the use of the Quell for persons with chronic musculoskeletal low back pain. The investigators hypothesize that those assigned to using the device will report reduced back pain compared with those in the control condition; with those using the device also showing improvement in sleep, mood, and level of activity. The investigators hypothesize that frequency of using the Quell (increased tolerability and adherence) will be correlated with greater reduction in pain. The investigators hypothesize that the device will be safe to use and will demonstrate a reduction in healthcare utilization (reduced clinic and Emergency Department visits). Finally, based on preliminary analyses limited by few subject numbers, the investigators will investigate whether certain individuals report greater benefit from using the Quell than others and, in particular, would predict that those with more intense and longer duration of pain will demonstrate most benefit.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be adults age 21 or older and diagnosed with axial musculoskeletal back pain without radiculopathy.
* Patients will be invited to participate if they own a smart phone (iPhone or Android device) and are able to download the pain app and the Quell Relief program app onto their device.
* Patients will also be included if they:

  1. have chronic pain for > 3 months' duration
  2. average 4 or greater on a pain intensity scale of 0 to 10
  3. are able to speak and understand English.

Exclusion Criteria:

* Patients will be excluded from participation if they meet any of the following criteria:

  1. diagnosis of cancer or any other malignant disease
  2. acute osteomyelitis or acute bone disease
  3. present or past Diagnostic and Statistical Manual-V diagnosis of schizophrenia, delusional disorder, psychotic disorder, or dissociative disorder that would be judged to interfere with study participation
  4. pregnancy
  5. any clinically unstable systemic illness judged to interfere with treatment
  6. a pain condition requiring urgent surgery
  7. an active substance use disorder, such as cocaine or IV heroin use, (positive on the Mini International Neuropsychiatric Interview; M.I.N.I. v.5.0) that would interfere with study participation
  8. any prescription opioid use for pain
  9. have an implanted cardiac pacemaker, defibrillator, or other implanted device. All subjects will be asked to not change their treatment during the study period.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

REFERENCES:
- [Result] Jamison RN, Wan L, Edwards RR, Mei A, Ross EL. Outcome of a High-Frequency Transcutaneous Electrical Nerve Stimulator (hfTENS) Device for Low Back Pain: A Randomized Controlled Trial. Pain Pract. 2019 Jun;19(5):466-475. doi: 10.1111/papr.12764. Epub 2019 Feb 4. PMID 30636101

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Subjects will receive the Quell device at the baseline visit and will be asked to use the device every day for 3 months.
- Control: Subjects will not receive the Quell device at the baseline visit, but they will receive one after 3 months.
Period: Overall Study
Arm/Group | Experimental | Control
Started | 35 | 33
Completed | 31 | 32
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Subjects will receive the Quell device
  Quell
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (14) | 45 (11) | 47 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 41
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 34 | 31 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 28 | 25 | 53
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Pain Duration [Mean (Standard Deviation); unit: years] | 12.5 (10.6) | 13.9 (13.4) | 13.2 (11.9)
Pain Average [Mean (Standard Deviation); unit: units on a scale] — Average pain score on a scale of 0-10, where 0 is no pain and 10 is worst possible pain. Higher value means worse pain representing a worse outcome.
  units on a scale | 5.2 (1.7) | 5.7 (1.4) | 5.5 (1.6)
Weight [Mean (Standard Deviation); unit: lbs] | 186.5 (60.0) | 175.0 (51.9) | 182.7 (51.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (6.0) | 30.7 (8.5) | 30.4 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity (Average)
Description: Rate average pain intensity using visual analog scale on a scale of 0-10, where 0 is no pain and 10 is worst possible pain. Higher scores mean a worse outcome.
Time Frame: 3 months
Population: For the experimental group, 35 subjects were consented, 4 subjects dropped out, 2 subjects did not complete the 3-month questionnaire, so 29 subjects were analyzed. For the control group, 33 subjects were consented, 1 subject dropped out, 1 subject did not complete the 3-month questionnaire, so 31 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 29 | 31
score on a scale | 4.0 (2.5) | 5.7 (1.9)

2. Primary Outcome: Average Pain Interference
Description: This measures the average pain interference with general activity, mood, walking ability, normal work, relations with others, sleep and enjoyment of life using visual analogue scale. On a scale of 0-10, 0 is no interference and 10 is extreme interference. Higher scores mean worse outcome.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 29 | 31
score on a scale | 3.2 (3.0) | 5.4 (2.3)

3. Primary Outcome: Pain Disability Index
Description: The Pain Disability Index (PDI) a simple and rapid instrument for measuring the impact that pain has on the ability of a person to participate in essential life activities. For each of the 7 categories of life activity listed, a score of 0 means no disability at all, and a score of 10 signifies that all of the activities in which you would normally be involved have been totally disrupted or prevented by your pain. The minimal index is 0 and maximal index is 70. The higher the index the greater the person's disability due to pain meaning a worse outcome.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 29 | 31
score on a scale | 26.3 (19.0) | 34.9 (16.7)

4. Primary Outcome: Pain Catastrophizing Scale
Description: Pain Catastrophizing Scale (PCS) has thirteen statements describing different thoughts and feelings that may be associated with pain. Using a 5-point scale from 0 (Not at all) to 4 (all the time), people indicate the degree to which they have these thoughts and feelings when they are experiencing pain. The sum has a minimum of 0 and a maximum of 52. Higher scores mean high levels of pain catastrophizing and worse outcome.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 29 | 31
score on a scale | 13.9 (12.6) | 25.1 (13.8)

5. Primary Outcome: Hospital Anxiety and Depression Scale Total Score
Description: Hospital Anxiety and Depression Scale (HADS) is commonly used to determine the levels of anxiety and depression that a person is experiencing. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. This outcome is a total score, which was calculated by adding the anxiety score and the depression score. Total score ranges from 0-42, with higher scores indicating a worse outcome.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 29 | 31
score on a scale | 15.2 (8.8) | 16.6 (7.6)

6. Secondary Outcome: Post-study Helpfulness Questionnaire
Description: The questionnaire asked the participants to rate how helpful was the device for the low back pain on a scale of 0-10. 0 is not helpful at all and 10 is very helpful. Higher value means better outcome.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 29 | 31
score on a scale | 4.7 (3.4) | NA (NA) — For the control group, the subjects received the device after they completed study, so they could not complete the 3-month helpfulness questionnaire.

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

LIMITATIONS AND CAVEATS:
1. followed for only three months
2. no active comparator treatment in the control group
3. hard to know how other treatments or environmental factors might have affected the outcome of this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02944513/Prot_SAP_001.pdf